CLINICAL TRIAL: NCT07271316
Title: Birth Control Supplement Study
Brief Title: Alii Supplement Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Sarah Hill, Professor, Texas Christian University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB#2025-383
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Nutrient Deficiency; Happiness; Digestive Health; Vulnerability to Disease; Mood Swings; Energy
Keywords: Hormonal Birth Control; Nutritional Depletion; Dietary Supplement

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The primary investigator and co-investigator will have knowledge as to what group each participant is in. However, the research assistants who will be the only individuals interacting with the participants will not have knowledge as to what group each participant is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Half of the participants will be randomly assigned by researchers to take a placebo. The researchers who are giving the participant the placebo will not know if they are giving the participant a placebo or the supplement. The placebo being used is the Magic Bullet Placebo Pill. Participants will take 3 placebo pills per day for 28 days.
  Interventions: Other: Placebo
- Alii Supplement (Experimental): Half of the participants will be randomly assigned by researchers to take the Alii Supplement. The investigators who are giving the participant the Alii supplement will not know if the participants are receiving a placebo or the supplement. Participants will take 3 pills per day for 28 days.
  Interventions: Dietary Supplement: Alii Supplement

INTERVENTIONS:
Dietary Supplement: Alii Supplement — This is the experimental group, looking to see how a supplement aiming to improve nutrition levels in hormonal birth control users may improve symptoms related to nutritional depletion. Per serving (3 capsules), the supplement contains 90 mg of Vitamin C, 25 μg of Vitamin D3, 135 mg of Vitamin E, 100 mg of Vitamin B1, 50 mg of Vitamin B2, 50mg of Vitamin B3, 50 mg of Vitamin B6, 567 μg DFE of Folate, 250 μg of Vitamin B12, 20mg of Pantothenic Acid, 100mg of Magnesium, 11mg of Zinc, 200 μg of Selenium, 300 mg of Tributyrin, and 50 mg of Coenzyme Q 10. The supplement also contains Hypromellose, Silicon Dioxide, Microcrystalline Cellulose, Magnesium Stearate, and Stearic Acid.
  Arms: Alii Supplement
Other: Placebo — This is the control group, so that the investigators can compare potential effects of the Alii supplement to the control group. The placebo contains Hypromellose and Microcrystalline Cellulose
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if the Alii Supplement can be used to reduce symptoms related to nutritional depletion in hormonal birth control pill users. The main questions it aims to answer are:

Does usage of the supplement increase happiness, decrease perceived vulnerability to disease, increase digestive health, decrease mood swings, and increase energy?

The investigators will compare the Alii Supplement to a placebo (a capsule that contains no drug) to see if the Alii Supplement works to reduce symptoms associated with nutritional depletion.

Participants will:

Take the placebo or Alii Supplement everyday for 28 days and visit the research office twice to fill out an online survey comprising of items examining the main outcome measures.

DETAILED DESCRIPTION:
This randomized, double-blind clinical trial will look to examine the efficacy of the Alii supplement, compared to a placebo, on reducing symptoms related to nutritional depletion in hormonal birth control pill users. This clinical trial will be conducted on 68 female university students. Participants will fill out measures of happiness, mood swings, digestive health, vulnerability to disease, and energy at time 1. Participants will then be randomly assigned to take a placebo or the Alii supplement for 28 days. Specifically, participants will take three capsules per day, with or without food. Participants will receive daily reminders to take their capsules. After taking the placebo or the supplement for 28 days, participants will again fill out the same measures of happiness, mood swings, digestive health, vulnerability to disease, and energy. Differences in these outcomes over time will be assessed to determine if taking the Alii supplement can improve these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be on the hormonal birth control pill as the investigators are testing the effectiveness of a supplement for women who take the hormonal birth control pill
* Participants must be willing to complete a follow up survey as this study will be multiple parts
* Participants must be willing to take a daily supplement as this study is testing how a supplement influences a variety of psychological outcomes
* Participants must be on the hormonal birth control pill for at least six months as participants who have been on the pill for less than 6 months may not be experiencing nutritional depletion yet
* If the investigators are able to do so, the investigators will only recruit participants who take the one-month hormonal birth control pill rather than the three month hormonal birth control pill, as the investigators are going to have participants come in after 28 days (day 2 of pack 1 and day 2 of pack 2) and participants on the three-month HBC pill may be on a 21 day cycle.
* Participants must have no food or medication allergies that will prevent the participants from safely taking the supplement
* Participants must not be taking any vitamins or participant must report willingness to abstain from taking vitamins during the study as individuals who are already taking vitamins may not be experiencing nutritional depletion associated with hormonal birth control
* If the investigators have the ability to do so, the investigators will only recruit participants who are not taking medications. Participants on various medications (e.g., SSRIs, ADHD medications, etc.) may report differing psychological states due to their medications, rather than the supplement. Therefore, it would be best to exclude those individuals if possible.

Exclusion Criteria:

* Participants cannot be naturally cycling as the investigators are testing a supplement for women on hormonal birth control
* Participants cannot be unwilling to complete a follow up study because this is a multi-part study
* Participants cannot be unwilling to take a supplement because the study centers around taking a supplement
* Participants cannot be on the hormonal birth control pill for less than 6 months as participants who have been on the pill for less than 6 months may not be experiencing nutritional depletion yet
* If the investigators are able to do so, participants cannot take the three month hormonal birth control pill, as the investigators are going to have participants come in after 28 days (day 2 of pack 1 and day 2 of pack 2) and participants on the three-month HBC pill may be on a 21 day cycle.
* Participants cannot have any food or medication allergies that will prevent the participants from safely taking the supplement
* Participants must not be taking any vitamins or participants must report willingness to abstain from taking vitamins during the study as individuals who are already taking vitamins may not be experiencing nutritional depletion associated with hormonal birth control
* If the investigators have the ability to do so, the investigators will only recruit participants who are not taking medications. Participants on various medications (e.g., SSRIs, ADHD medications, etc.) may report differing psychological states due to their medications, rather than the supplement. Therefore, it would be best to exclude those individuals if possible.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Levels of Perceived Vulnerability to Disease Scale after 1 Month of Drug Usage | From day 1 of supplement usage to the end of treatment at 4 weeks.
  Participants complete the Perceived Infectability Subscale (Duncan et al., 2009). For each scale item, 1 = Strongly disagree to 7 = Strongly agree. Higher scores indicate a higher perceived vulnerability to disease.
Change from Baseline in Levels of Happiness after 1 Month of Drug Usage | From day 1 of supplement usage to the end of treatment at 4 weeks.
  Participants complete the Short Depression-Happiness Scale (Joseph et al., 2004). For each scale item, 1 = Never... 4 = Often. Higher scores indicate higher levels of happiness.
Change from Baseline in Levels of Digestive Health after 1 Month of Drug Usage | From day 1 of supplement usage to the end of treatment at 4 weeks.
  Participants complete a modified version of the Birmingham IBS Symptom Questionnaire (Roalfe et al., 2008). For each scale item, 1: All of the time... 6: None of the time. Higher scores indicate better digestive health.
Change from Baseline in Levels of Mood Swings after 1 Month of Drug Usage | From day 1 of supplement usage to the end of treatment at 4 weeks.
  Participants complete the Modified Version of the Mood Instability Questionnaire-Trait (Yoon et al., 2021). For each scale item, 0 = not at all true, 1 = hardly true, 2 = moderately true, and 3 = exactly true. Higher scores indicate more mood swings.
Change from Baseline in Levels of Energy after 1 Month of Drug Usage | From day 1 of supplement usage to the end of treatment at 4 weeks.
  Participants complete the Multidimensional Fatigue Inventory (General Fatigue and Physical Fatigue Subscales; Smets et al., 1995). For each scale item, 1 = Yes, that is true... 5 = No, that is not true. Higher scores indicate higher energy levels.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Hill, PhD, Principal Investigator — Texas Christian University
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared either via OSF or upon request once the manuscript has been published. All data will be de-identified prior to sharing with other researchers. Supporting information (e.g., study protocol, informed consent forms, etc.) may be made available upon request. No time frame has been determined for length of time data are available.

REFERENCES:
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] Joseph S, Linley PA, Harwood J, Lewis CA, McCollam P. Rapid assessment of well-being: The Short Depression-Happiness Scale (SDHS). Psychol Psychother. 2004 Dec;77(Pt 4):463-78. doi: 10.1348/1476083042555406. PMID 15588455
- [Background] Yoon J, Ha TH, Oh S, Park YS, Ryoo HA, Yu HA, Hong SJ, Cho N, Lee CW, Jang Y, Lee W, Kim YR, Park KH, Park J, Park JY, Myung W. Development and Validation of the Mood Instability Questionnaire-Trait (MIQ-T). Medicina (Kaunas). 2021 Aug 18;57(8):838. doi: 10.3390/medicina57080838. PMID 34441044